CLINICAL TRIAL: NCT05803746
Title: PD-L2 Targeting Nanobody Radiotracer for PET Imaging of Solid Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022KT114
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Colorectal Cancer
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All enrolled participants will be allocated to this arm (single-arm study). Study participants will undergo 68Ga-Mirc415 PET/CT scan.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/ CT scan.

SUMMARY:
The objective of this study is to construct a noninvasive approach using 68Ga- Mirc415 PET/CT to detect the PD-L2 expression of tumor lesion in patients with colorectal cancer, lung cancer and other solid tumor to identify patients benefiting from anti-PD-(L)1 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75, male and female, with ECOG score of 0 or 1;
2. Subjects with head and neck tumors, lung cancer, esophageal cancer, breast cancer, ovarian cancer, cholangiocarcinoma, colorectal cancer, gastric cancer, pancreatic cancer, melanoma, bone or soft tissue sarcoma, solid tumors or suspected tumor subjects who intend to undergo pathological tissue biopsy or receive tumor surgical treatment in the near future (within 2 months);
3. The expected survival was more than 26 weeks;
4. Blood routine test, liver and kidney function meet the following standards: blood routine: WBC >= 4.0 x 10^9/L or neutrophil >= 1.5 x 10^9/:, PLT >= 100 x 10^9 / L, Hb >= 90g / L; Pt or APTT <= 1.5 upper limit of normal value; liver and kidney function: total bilirubin <= 1.5 x ULT (upper limit of normal value), ALT / AST <= 2.5 upper limit of normal value or <= 5 x ULT (subject with liver metastasis), ALP <= 2.5 upper limit of normal value (if bone metastasis or liver metastasis exists, ALP <= 4.5 upper limit of normal value); BUN <= 1.5 x ULT, SCR <= 1.5 x ULT;
5. According to RECIST1.1, there was at least one measurable target lesion;
6. Women must take effective contraceptive measures during the study period and within 6 months after the end of the study; men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period;
7. Understand and sign informed consent voluntarily with good compliance.

Exclusion Criteria:

1. The function of liver and kidney was seriously abnormal;
2. Preparation for pregnant, pregnant and lactating women;
3. Inability to lie flat for half an hour;
4. Suffering from claustrophobia or other mental disorders; 5) Other researchers considered it unsuitable to participate in the trial. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
MPR | [Time Frame: After 2-4 cycles of immunotherapy (each cycle is 28 days)]
  In the surgical pathology after neo-adjuvant immunotherapy, the proportion of active tumors was less than 10%.

SECONDARY OUTCOMES:
PFS | 2 years
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China